CLINICAL TRIAL: NCT01918124
Title: A Phase II Clinical Trial of Adjuvant Postoperative Irradiation Combined With Paclitaxel/Carboplatin(TP) or Cisplatin/Doxorubicin/Cyclophosphamide (CAP) Chemotherapy for Patients With High-risk Endometrial Cancer
Brief Title: A Phase II Trial of Adjuvant Radiotherapy Combined With Chemotherapy for Patients With High-risk Endometrial Cancer
Acronym: EC-0701
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fan Ming (Other)
Responsible Party: Sponsor-Investigator, Fan Ming, Shanghai Cancer Center, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070148-7
Record Dates: First submitted 2013-07-29; First posted 2013-08-07 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Prosthesis Survival
Keywords: disease free survival, overall survival
MeSH Terms: conditions — Prosthesis Failure | interventions — Radiotherapy; Cisplatin; Doxorubicin; Cyclophosphamide; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy combined with chemotherapy (Experimental): Arm Label: radiotherapy combined with chemotherapy:
  Radiotherapy:
  Pelvic radiation to 45 Gy, 1.8 Gy per day, five days per week (25 fractions) or intensive modulated pelvic radiotherapy, with brachytherapy boost to the vagina if total abdominal hysterectomy and bilateral salpingo-oophorectomy was done in surgery, or with paraaortic radiation if paraaortic lymphnode metastases were found after surgery.
  Cisplatin:
  Two courses cisplatin (50mg/m2) given on days 1 and 28 during radiotherapy.
  Cisplatin and Doxorubicin and Cyclophosphamide： Four courses of cisplatin (50mg/m2) and doxorubicin (60mg/m2) and cyclophosphamide (600mg/m2) given at 3 week intervals following completion of radiotherapy.
  Paclitaxel and Carboplatin： Or four courses of Paclitaxel(135mg/m2) and carboplatin (AUC=5) given at 3 week intervals following completion of radiotherapy.
  Interventions: Radiation: radiotherapy; Drug: Cisplatin; Drug: Cisplatin and Doxorubicin and Cyclophosphamide; Drug: Paclitaxel and Carboplatin

INTERVENTIONS:
Radiation: radiotherapy — Pelvic radiation to 45 Gy, 1.8 Gy per day, five days per week (25 fractions) or intensive modulated pelvic radiotherapy, with brachytherapy boost to the vagina if total abdominal hysterectomy and bilateral salpingo-oophorectomy was done in surgery, or with paraaortic radiation if paraaortic lymphnode metastases were found after surgery.
Drug: Cisplatin — Two courses cisplatin (50mg/m2) given on days 1 and 28 during radiotherapy.
Drug: Cisplatin and Doxorubicin and Cyclophosphamide — Four courses of cisplatin (50mg/m2) and doxorubicin (60mg/m2) and cyclophosphamide (600mg/m2) chemotherapy given at 3 week intervals following completion of radiotherapy.
Drug: Paclitaxel and Carboplatin — Or four courses of Paclitaxel(135mg/m2) and carboplatin (AUC=5) given at 3 week intervals following completion of radiotherapy.

SUMMARY:
This phase II clinical trial was designed to assess the feasibility, safety, toxicity, recurrence and survival pattern when TP or CAP chemotherapy was combined with adjuvant radiation for patients with high-risk endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a hysterectomy (total abdominal, vaginal hysterectomy, or laparoscopic-assisted vaginal hysterectomy) or modified radical hysterectomy or radical hysterectomy and bilateral salpingo-oophorectomy no more than 8 weeks prior to start of radiation therapy.

Additional surgical staging procedures are permissible but not required.

* Risk factors: patients must fit one of the following:

  * Pelvic lymph node metastases
  * Paraaortic lymph node metastases
  * Grade 3 with myometrial invasion >50%
  * With stromal invasion of cervix
  * Known extrauterine disease (excluding second primary) confined to the pelvis.
  * High risk pathological type include: uterine papillary serous carcinoma, clear cell carcinoma, squamous cell carcinoma, undifferentiated carcinoma,
* No known gross residual disease, or distant metastases.
* Eastern Cooperative Oncology Group (ECOG) score<=2; Age 18~75.
* White Blood Cell (WBC)≥4000/mm3, granulocytes ≥1500/mcl, platelets≥100,000/mcl.
* Acceptable hepatic and renal function: creatinine <=1.4 mg%, bilirubin and serum glutamate oxaloacetate transaminase (SGOT) <=2*normal.
* No medical contraindications to chemotherapy, or radiation therapy.
* Study-specific signed informed consent.

Exclusion Criteria:

* Prior pelvic radiation therapy.
* Positive peritoneal cytology only for stage IIIa (FIGO 1998).
* With history of other malignancies less than 5 years.
* With gross residual disease, or distant metastases.
* With endometrioid endometrial carcinoma and no risk factors:

  * with myometrial invasion <50%
  * Grade 1~2, with myometrial invasion >50%
* With serious internal diseases which affect designed treatment
* With psychotic disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival(DFS) | From date of randomization until the date of first documented progression, assedded up to 60 months
  From date of randomization until the date of first documented progression, assessed up to 60 months.

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of randomization until the date of death from any cause, assedded up to 60 months.
  From date of randomization until the date of death from any cause, assessed up to 60 months.

OTHER OUTCOMES:
Number of patients with adverse events and number of patients completed the treatments | up to 5 years
  Number of patients completed the treatment and number of patients with adverse events up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Huaying Wang, Doctor, Study Chair — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Ren Y, Huang X, Shan B, Wu X, Huang X, Shi D, Wang H. Adjuvant concurrent chemoradiation followed by chemotherapy for high-risk endometrial cancer. Gynecol Oncol. 2016 Jan;140(1):58-63. doi: 10.1016/j.ygyno.2015.11.021. Epub 2015 Nov 24. PMID 26607778
- See also: Related Info — http://www.shca.org.cn